CLINICAL TRIAL: NCT03826667
Title: Post-market Clinical Follow-up (PMCF) Study on PEEK Suture Anchors for Shoulder Indications
Brief Title: PMCF Study on PEEK Suture Anchors for Shoulder Indications
Status: Completed | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018.16.SMD.PEEK.RET.SHD
Record Dates: First submitted 2019-01-30; First posted 2019-02-01 (Actual); Results first posted 2022-04-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-02

CONDITIONS: Soft Tissue to Bone Fixation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Polyetheretherketone (PEEK) Shoulder Suture Anchors — PEEK Suture Anchors, which include:
  * HEALICOIL™ PK Preloaded Suture Anchors
  * BIORAPTOR™ 2.3 PK Suture Anchors/BIORAPTOR™ Curved 2.3 PK Suture Anchors
  * BIORAPTOR™ Knotless Suture Anchors
  * MULTIFIX™ S Ultra Knotless Fixation System
  * FOOTPRINT™ Ultra PK Suture Anchors
  * TWINFIX™ Ultra PK Suture Anchors/TWINFIX™ Ultra Preloaded and with Needles
  * SPEEDSCREW™ Knotless Fixation System
  * SpeedLock Knotless Fixation Device

SUMMARY:
Post-market clinical follow-up on the PEEK Suture Anchors in the shoulder.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have undergone shoulder joint repair using the study devices.
2. Subjects aged 18 years and older at the time of surgery.

Exclusion Criteria:

1. Subjects who are < 12 months post-operative.
2. Subject is entered in another investigational drug, biologic, or device study or has been treated with an investigational product within 30 days prior to surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have received PEEK Suture Anchors implanted in the shoulder
Sampling Method: Non-Probability Sample
Enrollment: 464 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2019-08-28 (Actual); Study Completion 2019-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judth Horner, Study Chair — Smith & Nephew, Inc.
Locations (11):
- United States (11):
  - Grandview Medical Center, Birmingham, Alabama
  - OrthoArizona, Phoenix, Arizona
  - University of Colorado- Denver, Denver, Colorado
  - Holy Cross Hospital/Orthopedic Institute, Fort Lauderdale, Florida
  - OrthoAtlanta, Lawrenceville, Georgia
  - Community Hospital, Oklahoma City, Oklahoma
  - University Orthopedics Center, Altoona, Pennsylvania
  - Houston Methodist at Baytown, Baytown, Texas
  - Texas Orthopedic Hospital - Houston, Houston, Texas
  - Aspen Orthopedics at New Berlin, New Berlin, Wisconsin
  - Aspen Orthopedics at West Allis, West Allis, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: It was intended to enroll participants for 8 PEEK suture anchor devices; however, no participants were enrolled for the BIORAPTOR™ Knotless Suture Anchors, resulting in 7 suture anchor groups being analyzed. A total of 464 participants were enrolled in the study and 467 joints were observed. Multiple devices were implanted in 124 participants.
Units Other Than Participants: joints
Groups:
- Polyetheretherketone (PEEK) Shoulder Suture Anchors: Participants who have received PEEK Suture Anchors in the shoulder which included:
  HEALICOIL™ PK Preloaded Suture Anchors, BIORAPTOR™ 2.3 PK Suture Anchors/BIORAPTOR™ Curved 2.3 PK Suture Anchors, MULTIFIX™ S Ultra Knotless Fixation System, FOOTPRINT™ Ultra PK Suture Anchors, TWINFIX™ Ultra PK Suture Anchors/TWINFIX™ Ultra Preloaded and with Needles, SPEEDSCREW™ Knotless Fixation System, SpeedLock Knotless Fixation Device
Period: Overall Study
Arm/Group | Polyetheretherketone (PEEK) Shoulder Suture Anchors
Started | 464; 467 joints
HEALICOIL™ PK Preloaded Suture Anchors (Type of suture anchor received at start) | 193; 193 joints
BIORAPTOR™ 2.3 PK Suture Anchors/BIORAPTOR™ Curved 2.3 PK Suture Anchors (Type of suture anchor received at start) | 41; 41 joints
MULTIFIX™ S Ultra Knotless Fixation System (Type of suture anchor received at start) | 78; 78 joints
FOOTPRINT™ Ultra PK Suture Anchors (Type of suture anchor received at start) | 136; 138 joints
TWINFIX™ Ultra PK Suture Anchors/TWINFIX™ Ultra Preloaded and With Needles (Type of suture anchor received at start) | 57; 57 joints
SPEEDSCREW™ Knotless Fixation System (Type of suture anchor received at start) | 59; 59 joints
SpeedLock Knotless Fixation Device (Type of suture anchor received at start) | 18; 18 joints
Completed | 443; 446 joints
Not Completed | 21; 21 joints
Not completed — Protocol deviation | 21

BASELINE CHARACTERISTICS:
Population: Participants enrolled in the study who had previously undergone shoulder repair using PEEK suture anchors (i.e., retrospective data). The type(s) of PEEK anchor used during surgery was surgeon decision on a case by case basis. Multiple anchor types could be used in one surgery if required. 124 participants had multiple devices implanted. Participants with bilateral surgeries had both surgeries recorded independently. Device data analyzed individually dependent on unique suture anchor implanted.
Units Other Than Participants: joints
Arm/Group | Polyetheretherketone (PEEK) Shoulder Suture Anchors
Number analyzed (Participants) | 464
Number analyzed (joints) | 467
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.00 (14.10)
Sex: Female, Male [Count of Units; unit: joints]
  Female | 190
  Male | 277
Ethnicity (NIH/OMB) [Count of Units; unit: joints]
  Hispanic or Latino | 30
  Not Hispanic or Latino | 367
  Unknown or Not Reported | 70
Race/Ethnicity, Customized [Count of Units; unit: joints]
  American Indian or Alaska Native: No | 462
  American Indian or Alaska Native: Yes | 5
  Asian: No | 464
  Asian: Yes | 3
  Black or African American: No | 444
  Black or African American: Yes | 23
  Native Hawaiian or Other Pacific Islander: No | 465
  Native Hawaiian or Other Pacific Islander: Yes | 2
  White: No | 94
  White: Yes | 373
  Other: No | 403
  Other: Yes | 64
Region of Enrollment [Number; unit: joints]
  United States | 467
Location of Device Implantation [Count of Units; unit: joints]
  Left Shoulder | 194
  Right Shoulder | 271
  Bilaterally | 2
Duration of Surgery [Mean (Standard Deviation); unit: minutes] — Population: Data was not available for all participants due to the retrospective nature of the study.
  minutes
    number analyzed (Participants) | 113
    (all) | 99.2 (50.7)
Duration of time from injury to surgery [Mean (Standard Deviation); unit: days] — Population: Data not available for all participants due to the retrospective nature of the study.
  days
    number analyzed (Participants) | 235
    (all) | 405.7 (929.2)
Any Medical History [Count of Units; unit: joints]
  Yes | 392
  No | 75
Number of Participant Joints Treated by Indication [Count of Units; unit: joints]
  Bankart lesion repair | 12
  SLAP lesion repair | 2
  Capsular shift | 5
  Rotator cuff repair | 413
  Biceps tenodesis | 33
  Other | 2
Disposition of Suture Anchors [Count of Participants; unit: Participants] — Count of participants by unique PEEK Suture Anchors implanted. Population: Information provided based on the unique device implanted. Out of 464 overall participants, 124 were implanted with multiple Suture Anchors (devices).
  Participants
    HEALICOIL™ PK Preloaded Suture Anchors | 193
    BIORAPTOR™ 2.3 PK Suture Anchor / BIORAPTOR™ Curved 2.3 PK Suture Anchor | 41
    MULTIFIX™ S Ultra Knotless Fixation System | 78
    FOOTPRINT™ Ultra PK Suture Anchor | 136
    TWINFIX™ Ultra PK Suture Anchor | 57
    SPEEDSCREW™ Knotless Fixation System | 59
    SpeedLock Knotless Fixation Device | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Success of the Study Devices in the Shoulder Over a Time Period of 6 Months After Intervention
Description: Clinical success was defined as shoulder repairs without signs of device failure and/or re-intervention as assessed by the surgeon. Specifically, clinical success was considered "Yes" based on the following 3 main criteria:
  * no inflammatory or allergic response
  * no device-related adverse event (AE)
  * no device deficiencies (DDs) leading to revision surgery (re intervention) on the index shoulder
Time Frame: 6 months
Population: Number of participants analyzed at the specified time frame for each row indicates participant provided retrospective data for the PEEK Suture Anchor identified. Some participants were implanted with multiple Suture Anchors (devices).Data was analyzed independently based on specific device implanted (i.e., participants with multiple devices were analyzed individually by unique suture anchor). Overall number of participants analyzed indicates combined total of distinct participants assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Polyetheretherketone (PEEK) Shoulder Suture Anchors
Number analyzed (Participants) | 458
Participants
  HEALICOIL™ PK Preloaded Suture Anchors: number analyzed (Participants) | 191
  HEALICOIL™ PK Preloaded Suture Anchors: Yes | 185
  HEALICOIL™ PK Preloaded Suture Anchors: No | 6
  BIORAPTOR™ 2.3 PK Suture Anchor / BIORAPTOR™ Curved 2.3 PK Suture Anchor: number analyzed (Participants) | 41
  BIORAPTOR™ 2.3 PK Suture Anchor / BIORAPTOR™ Curved 2.3 PK Suture Anchor: Yes | 38
  BIORAPTOR™ 2.3 PK Suture Anchor / BIORAPTOR™ Curved 2.3 PK Suture Anchor: No | 3
  MULTIFIX™ S Ultra Knotless Fixation System: number analyzed (Participants) | 77
  MULTIFIX™ S Ultra Knotless Fixation System: Yes | 71
  MULTIFIX™ S Ultra Knotless Fixation System: No | 6
  FOOTPRINT™ Ultra PK Suture Anchor: number analyzed (Participants) | 131
  FOOTPRINT™ Ultra PK Suture Anchor: Yes | 128
  FOOTPRINT™ Ultra PK Suture Anchor: No | 3
  TWINFIX™ Ultra PK Suture Anchor: number analyzed (Participants) | 57
  TWINFIX™ Ultra PK Suture Anchor: Yes | 57
  TWINFIX™ Ultra PK Suture Anchor: No | 0
  SPEEDSCREW™ Knotless Fixation System: number analyzed (Participants) | 59
  SPEEDSCREW™ Knotless Fixation System: Yes | 58
  SPEEDSCREW™ Knotless Fixation System: No | 1
  SpeedLock Knotless Fixation Device: number analyzed (Participants) | 18
  SpeedLock Knotless Fixation Device: Yes | 18
  SpeedLock Knotless Fixation Device: No | 0

2. Secondary Outcome: Number of Participants With Clinical Success of the Study Devices in the Shoulder Over a Time Period of 12 Months After Intervention
Description: as for outcome 1
Time Frame: 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Polyetheretherketone (PEEK) Shoulder Suture Anchors
Number analyzed (Participants) | 85
Participants
  HEALICOIL™ PK Preloaded Suture Anchors: number analyzed (Participants) | 51
  HEALICOIL™ PK Preloaded Suture Anchors: Yes | 50
  HEALICOIL™ PK Preloaded Suture Anchors: No | 1
  BIORAPTOR™ 2.3 PK Suture Anchor / BIORAPTOR™ Curved 2.3 PK Suture Anchor: number analyzed (Participants) | 5
  BIORAPTOR™ 2.3 PK Suture Anchor / BIORAPTOR™ Curved 2.3 PK Suture Anchor: Yes | 5
  BIORAPTOR™ 2.3 PK Suture Anchor / BIORAPTOR™ Curved 2.3 PK Suture Anchor: No | 0
  MULTIFIX™ S Ultra Knotless Fixation System: number analyzed (Participants) | 18
  MULTIFIX™ S Ultra Knotless Fixation System: Yes | 17
  MULTIFIX™ S Ultra Knotless Fixation System: No | 1
  FOOTPRINT™ Ultra PK Suture Anchor: number analyzed (Participants) | 18
  FOOTPRINT™ Ultra PK Suture Anchor: Yes | 16
  FOOTPRINT™ Ultra PK Suture Anchor: No | 2
  TWINFIX™ Ultra PK Suture Anchor: number analyzed (Participants) | 6
  TWINFIX™ Ultra PK Suture Anchor: Yes | 6
  TWINFIX™ Ultra PK Suture Anchor: No | 0
  SPEEDSCREW™ Knotless Fixation System: number analyzed (Participants) | 5
  SPEEDSCREW™ Knotless Fixation System: Yes | 4
  SPEEDSCREW™ Knotless Fixation System: No | 1
  SpeedLock Knotless Fixation Device: number analyzed (Participants) | 2
  SpeedLock Knotless Fixation Device: Yes | 2
  SpeedLock Knotless Fixation Device: No | 0

3. Secondary Outcome: Visual Analog Scale (VAS) - Pain
Description: The VAS is a continuous scale comprised of a horizontal line 100 millimeters (mm) in length, anchored by 2 verbal descriptors, one for each symptom extreme. The VAS pain score is presented on a scale ranging from 0 to 10. A score of 0 represents no pain (0 mm) and a score of 10 indicates extreme/unbearable pain (100 mm). The VAS rating was recorded retrospectively, per standard of care at 6 and 12 months post-surgery.
Time Frame: 6 and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Polyetheretherketone (PEEK) Shoulder Suture Anchors
Number analyzed (Participants) | 100
score on a scale
  HEALICOIL™ PK Preloaded Suture Anchors: 6 months: number analyzed (Participants) | 77
  HEALICOIL™ PK Preloaded Suture Anchors: 6 months | 1.8 (2.1)
  HEALICOIL™ PK Preloaded Suture Anchors: 12 months: number analyzed (Participants) | 27
  HEALICOIL™ PK Preloaded Suture Anchors: 12 months | 2.4 (1.8)
  BIORAPTOR™ 2.3 PK Suture Anchor / BIORAPTOR™ Curved 2.3 PK Suture Anchor: 6 months: number analyzed (Participants) | 8
  BIORAPTOR™ 2.3 PK Suture Anchor / BIORAPTOR™ Curved 2.3 PK Suture Anchor: 6 months | 2.5 (2.8)
  BIORAPTOR™ 2.3 PK Suture Anchor / BIORAPTOR™ Curved 2.3 PK Suture Anchor: 12 months: number analyzed (Participants) | 2
  BIORAPTOR™ 2.3 PK Suture Anchor / BIORAPTOR™ Curved 2.3 PK Suture Anchor: 12 months | 4.5 (0.7)
  MULTIFIX™ S Ultra Knotless Fixation System: 6 months: number analyzed (Participants) | 47
  MULTIFIX™ S Ultra Knotless Fixation System: 6 months | 2.2 (2.1)
  MULTIFIX™ S Ultra Knotless Fixation System: 12 months: number analyzed (Participants) | 15
  MULTIFIX™ S Ultra Knotless Fixation System: 12 months | 2.3 (1.9)
  FOOTPRINT™ Ultra PK Suture Anchor: 6 months: number analyzed (Participants) | 3
  FOOTPRINT™ Ultra PK Suture Anchor: 6 months | 2.3 (2.1)
  FOOTPRINT™ Ultra PK Suture Anchor: 12 months: number analyzed (Participants) | 0
  TWINFIX™ Ultra PK Suture Anchor: 6 months: number analyzed (Participants) | 0
  TWINFIX™ Ultra PK Suture Anchor: 12 months: number analyzed (Participants) | 0
  SPEEDSCREW™ Knotless Fixation System: 6 months: number analyzed (Participants) | 5
  SPEEDSCREW™ Knotless Fixation System: 6 months | 1.4 (3.1)
  SPEEDSCREW™ Knotless Fixation System: 12 months: number analyzed (Participants) | 0
  SpeedLock Knotless Fixation Device: 6 months: number analyzed (Participants) | 4
  SpeedLock Knotless Fixation Device: 6 months | 0 (0)
  SpeedLock Knotless Fixation Device: 12 months: number analyzed (Participants) | 0

4. Secondary Outcome: Count of Participants With Range of Motion (ROM) Full Functional Arc
Description: Range of motion defined as the participant having a full functional arc "Yes" or "No" at 6 month and 12 month post-operative visits.
Time Frame: 6 and 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Polyetheretherketone (PEEK) Shoulder Suture Anchors
Number analyzed (Participants) | 348
Participants
  HEALICOIL™ PK Preloaded Suture Anchors: 6 months: number analyzed (Participants) | 163
  HEALICOIL™ PK Preloaded Suture Anchors: 6 months: Has full functional arc: Yes | 111
  HEALICOIL™ PK Preloaded Suture Anchors: 6 months: Has full functional arc: No | 48
  HEALICOIL™ PK Preloaded Suture Anchors: 6 months: Has full functional arc: Unknown | 4
  HEALICOIL™ PK Preloaded Suture Anchors: 12 months: number analyzed (Participants) | 49
  HEALICOIL™ PK Preloaded Suture Anchors: 12 months: Has full functional arc: Yes | 37
  HEALICOIL™ PK Preloaded Suture Anchors: 12 months: Has full functional arc: No | 10
  HEALICOIL™ PK Preloaded Suture Anchors: 12 months: Has full functional arc: Unknown | 2
  BIORAPTOR™ 2.3 PK Suture Anchor / BIORAPTOR™ Curved 2.3 PK Suture Anchor: 6 months: number analyzed (Participants) | 33
  BIORAPTOR™ 2.3 PK Suture Anchor / BIORAPTOR™ Curved 2.3 PK Suture Anchor: 6 months: Has full functional arc: Yes | 29
  BIORAPTOR™ 2.3 PK Suture Anchor / BIORAPTOR™ Curved 2.3 PK Suture Anchor: 6 months: Has full functional arc: No | 3
  BIORAPTOR™ 2.3 PK Suture Anchor / BIORAPTOR™ Curved 2.3 PK Suture Anchor: 6 months: Has full functional arc: Unknown | 1
  BIORAPTOR™ 2.3 PK Suture Anchor / BIORAPTOR™ Curved 2.3 PK Suture Anchor: 12 months: number analyzed (Participants) | 2
  BIORAPTOR™ 2.3 PK Suture Anchor / BIORAPTOR™ Curved 2.3 PK Suture Anchor: 12 months: Has full functional arc: Yes | 1
  BIORAPTOR™ 2.3 PK Suture Anchor / BIORAPTOR™ Curved 2.3 PK Suture Anchor: 12 months: Has full functional arc: No | 1
  BIORAPTOR™ 2.3 PK Suture Anchor / BIORAPTOR™ Curved 2.3 PK Suture Anchor: 12 months: Has full functional arc: Unknown | 0
  MULTIFIX™ S Ultra Knotless Fixation System: 6 months: number analyzed (Participants) | 51
  MULTIFIX™ S Ultra Knotless Fixation System: 6 months: Has full functional arc: Yes | 35
  MULTIFIX™ S Ultra Knotless Fixation System: 6 months: Has full functional arc: No | 12
  MULTIFIX™ S Ultra Knotless Fixation System: 6 months: Has full functional arc: Unknown | 4
  MULTIFIX™ S Ultra Knotless Fixation System: 12 months: number analyzed (Participants) | 16
  MULTIFIX™ S Ultra Knotless Fixation System: 12 months: Has full functional arc: Yes | 9
  MULTIFIX™ S Ultra Knotless Fixation System: 12 months: Has full functional arc: No | 7
  MULTIFIX™ S Ultra Knotless Fixation System: 12 months: Has full functional arc: Unknown | 0
  FOOTPRINT™ Ultra PK Suture Anchor: 6 months: number analyzed (Participants) | 105
  FOOTPRINT™ Ultra PK Suture Anchor: 6 months: Has full functional arc: Yes | 90
  FOOTPRINT™ Ultra PK Suture Anchor: 6 months: Has full functional arc: No | 14
  FOOTPRINT™ Ultra PK Suture Anchor: 6 months: Has full functional arc: Unknown | 1
  FOOTPRINT™ Ultra PK Suture Anchor: 12 months: number analyzed (Participants) | 19
  FOOTPRINT™ Ultra PK Suture Anchor: 12 months: Has full functional arc: Yes | 17
  FOOTPRINT™ Ultra PK Suture Anchor: 12 months: Has full functional arc: No | 2
  FOOTPRINT™ Ultra PK Suture Anchor: 12 months: Has full functional arc: Unknown | 0
  TWINFIX™ Ultra PK Suture Anchor: 6 months: number analyzed (Participants) | 0
  TWINFIX™ Ultra PK Suture Anchor: 12 months: number analyzed (Participants) | 0
  SPEEDSCREW™ Knotless Fixation System: 6 months: number analyzed (Participants) | 54
  SPEEDSCREW™ Knotless Fixation System: 6 months: Has full functional arc: Yes | 46
  SPEEDSCREW™ Knotless Fixation System: 6 months: Has full functional arc: No | 5
  SPEEDSCREW™ Knotless Fixation System: 6 months: Has full functional arc: Unknown | 3
  SPEEDSCREW™ Knotless Fixation System: 12 months: number analyzed (Participants) | 5
  SPEEDSCREW™ Knotless Fixation System: 12 months: Has full functional arc: Yes | 4
  SPEEDSCREW™ Knotless Fixation System: 12 months: Has full functional arc: No | 1
  SPEEDSCREW™ Knotless Fixation System: 12 months: Has full functional arc: Unknown | 0
  SpeedLock Knotless Fixation Device: 6 months: number analyzed (Participants) | 18
  SpeedLock Knotless Fixation Device: 6 months: Has full functional arc: Yes | 18
  SpeedLock Knotless Fixation Device: 6 months: Has full functional arc: No | 0
  SpeedLock Knotless Fixation Device: 6 months: Has full functional arc: Unknown | 0
  SpeedLock Knotless Fixation Device: 12 months: number analyzed (Participants) | 2
  SpeedLock Knotless Fixation Device: 12 months: Has full functional arc: Yes | 2
  SpeedLock Knotless Fixation Device: 12 months: Has full functional arc: No | 0
  SpeedLock Knotless Fixation Device: 12 months: Has full functional arc: Unknown | 0

5. Secondary Outcome: Range of Motion (ROM)
Description: Forward flexion angle, internal rotation angle, and external rotation angle captured in degrees based on physician's Standard of Care.
Time Frame: 6 and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Polyetheretherketone (PEEK) Shoulder Suture Anchors
Number analyzed (Participants) | 70
degrees
  HEALICOIL™ PK Preloaded Suture Anchors: Forward Flexion Angle (6 months): number analyzed (Participants) | 45
  HEALICOIL™ PK Preloaded Suture Anchors: Forward Flexion Angle (6 months) | 157 (20.2)
  HEALICOIL™ PK Preloaded Suture Anchors: Internal Rotation Angle (6 months): number analyzed (Participants) | 6
  HEALICOIL™ PK Preloaded Suture Anchors: Internal Rotation Angle (6 months) | 25.7 (40.6)
  HEALICOIL™ PK Preloaded Suture Anchors: External Rotation (6 months): number analyzed (Participants) | 39
  HEALICOIL™ PK Preloaded Suture Anchors: External Rotation (6 months) | 49.3 (20.5)
  HEALICOIL™ PK Preloaded Suture Anchors Forward Flexion Angle (12 months): number analyzed (Participants) | 9
  HEALICOIL™ PK Preloaded Suture Anchors Forward Flexion Angle (12 months) | 141.1 (39.8)
  HEALICOIL™ PK Preloaded Suture Anchors Internal Rotation Angle (12 months): number analyzed (Participants) | 2
  HEALICOIL™ PK Preloaded Suture Anchors Internal Rotation Angle (12 months) | 75 (21.2)
  HEALICOIL™ PK Preloaded Suture Anchors External Rotation (12 months): number analyzed (Participants) | 8
  HEALICOIL™ PK Preloaded Suture Anchors External Rotation (12 months) | 59.4 (25.7)
  BIORAPTOR™ 2.3 PK /BIORAPTOR™ Curved 2.3 PK Suture Anchor: Forward Flexion Angle (6 months): number analyzed (Participants) | 2
  BIORAPTOR™ 2.3 PK /BIORAPTOR™ Curved 2.3 PK Suture Anchor: Forward Flexion Angle (6 months) | 89 (100.4)
  BIORAPTOR™ 2.3 PK /BIORAPTOR™ Curved 2.3 PK Suture Anchor: Internal Rotation Angle (6 months): number analyzed (Participants) | 3
  BIORAPTOR™ 2.3 PK /BIORAPTOR™ Curved 2.3 PK Suture Anchor: Internal Rotation Angle (6 months) | 60 (15)
  BIORAPTOR™ 2.3 PK /BIORAPTOR™ Curved 2.3 PK Suture Anchor: External Rotation (6 months): number analyzed (Participants) | 3
  BIORAPTOR™ 2.3 PK /BIORAPTOR™ Curved 2.3 PK Suture Anchor: External Rotation (6 months) | 100 (30)
  BIORAPTOR™ 2.3 PK /BIORAPTOR™ Curved 2.3 PK Suture Anchor: Forward Flexion Angle (12 months): number analyzed (Participants) | 0
  BIORAPTOR™ 2.3 PK /BIORAPTOR™ Curved 2.3 PK Suture Anchor: Internal Rotation Angle (12 months): number analyzed (Participants) | 0
  BIORAPTOR™ 2.3 PK /BIORAPTOR™ Curved 2.3 PK Suture Anchor: External Rotation (12 months): number analyzed (Participants) | 0
  MULTIFIX™ S Ultra Knotless Fixation System: Forward Flexion Angle (6 months): number analyzed (Participants) | 10
  MULTIFIX™ S Ultra Knotless Fixation System: Forward Flexion Angle (6 months) | 122.5 (39.4)
  MULTIFIX™ S Ultra Knotless Fixation System: Internal Rotation Angle (6 months): number analyzed (Participants) | 1
  MULTIFIX™ S Ultra Knotless Fixation System: Internal Rotation Angle (6 months) | 90 (NA) — Standard deviation not calculated whenever there was only 1 participant's data available
  MULTIFIX™ S Ultra Knotless Fixation System: External Rotation (6 months): number analyzed (Participants) | 5
  MULTIFIX™ S Ultra Knotless Fixation System: External Rotation (6 months) | 59.8 (25.3)
  MULTIFIX™ S Ultra Knotless Fixation System: Forward Flexion Angle (12 months): number analyzed (Participants) | 6
  MULTIFIX™ S Ultra Knotless Fixation System: Forward Flexion Angle (12 months) | 141.7 (38.2)
  MULTIFIX™ S Ultra Knotless Fixation System: Internal Rotation Angle (12 months): number analyzed (Participants) | 2
  MULTIFIX™ S Ultra Knotless Fixation System: Internal Rotation Angle (12 months) | 75 (21.2)
  MULTIFIX™ S Ultra Knotless Fixation System: External Rotation (12 months): number analyzed (Participants) | 5
  MULTIFIX™ S Ultra Knotless Fixation System: External Rotation (12 months) | 76 (21.9)
  FOOTPRINT™ Ultra PK Suture Anchor: Forward Flexion Angle (6 months): number analyzed (Participants) | 14
  FOOTPRINT™ Ultra PK Suture Anchor: Forward Flexion Angle (6 months) | 137.5 (35.9)
  FOOTPRINT™ Ultra PK Suture Anchor: Internal Rotation Angle (6 months): number analyzed (Participants) | 4
  FOOTPRINT™ Ultra PK Suture Anchor: Internal Rotation Angle (6 months) | 86.3 (30.9)
  FOOTPRINT™ Ultra PK Suture Anchor: External Rotation (6 months): number analyzed (Participants) | 14
  FOOTPRINT™ Ultra PK Suture Anchor: External Rotation (6 months) | 50 (22.7)
  FOOTPRINT™ Ultra PK Suture Anchor: Forward Flexion Angle (12 months): number analyzed (Participants) | 2
  FOOTPRINT™ Ultra PK Suture Anchor: Forward Flexion Angle (12 months) | 140 (28.3)
  FOOTPRINT™ Ultra PK Suture Anchor: Internal Rotation Angle (12 months): number analyzed (Participants) | 0
  FOOTPRINT™ Ultra PK Suture Anchor: External Rotation (12 months): number analyzed (Participants) | 2
  FOOTPRINT™ Ultra PK Suture Anchor: External Rotation (12 months) | 60 (0)
  TWINFIX™ Ultra PK Suture Anchor: Forward Flexion Angle (6 months): number analyzed (Participants) | 0
  TWINFIX™ Ultra PK Suture Anchor: Internal Rotation Angle (6 months): number analyzed (Participants) | 0
  TWINFIX™ Ultra PK Suture Anchor: External Rotation (6 months): number analyzed (Participants) | 0
  TWINFIX™ Ultra PK Suture Anchor: Forward Flexion Angle (12 months): number analyzed (Participants) | 0
  TWINFIX™ Ultra PK Suture Anchor: Internal Rotation Angle (12 months): number analyzed (Participants) | 0
  TWINFIX™ Ultra PK Suture Anchor: External Rotation (12 months): number analyzed (Participants) | 0
  SPEEDSCREW™ Knotless Fixation System: Forward Flexion Angle (6 months): number analyzed (Participants) | 5
  SPEEDSCREW™ Knotless Fixation System: Forward Flexion Angle (6 months) | 122 (46.0)
  SPEEDSCREW™ Knotless Fixation System: Internal Rotation Angle (6 months): number analyzed (Participants) | 0
  SPEEDSCREW™ Knotless Fixation System: External Rotation (6 months): number analyzed (Participants) | 5
  SPEEDSCREW™ Knotless Fixation System: External Rotation (6 months) | 35 (10)
  SPEEDSCREW™ Knotless Fixation System: Forward Flexion Angle (12 months): number analyzed (Participants) | 1
  SPEEDSCREW™ Knotless Fixation System: Forward Flexion Angle (12 months) | 130 (NA) — Standard deviation not calculated whenever there was only 1 participant's data available
  SPEEDSCREW™ Knotless Fixation System: Internal Rotation Angle (12 months): number analyzed (Participants) | 0
  SPEEDSCREW™ Knotless Fixation System: External Rotation (12 months): number analyzed (Participants) | 1
  SPEEDSCREW™ Knotless Fixation System: External Rotation (12 months) | 50 (NA) — Standard deviation not calculated whenever there was only 1 participant's data available
  SpeedLock Knotless Fixation Device: Forward Flexion Angle (6 months): number analyzed (Participants) | 0
  SpeedLock Knotless Fixation Device: Internal Rotation Angle (6 months): number analyzed (Participants) | 0
  SpeedLock Knotless Fixation Device: External Rotation (6 months): number analyzed (Participants) | 0
  SpeedLock Knotless Fixation Device: Forward Flexion Angle (12 months): number analyzed (Participants) | 0
  SpeedLock Knotless Fixation Device: Internal Rotation Angle (12 months): number analyzed (Participants) | 0
  SpeedLock Knotless Fixation Device: External Rotation (12 months): number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Surgery to End of Study (EOS) visit, approximately 12 months
Description: AE reporting was collected retrospectively from the information available in the participant's medical records. A total of 464 participants were enrolled in the study. However, there were 124 participants with multiple devices implanted. Participant Suture Anchor data analyzed independently based on device implanted (i.e., participants implanted with multiple devices were analyzed individually based on unique suture anchor).
Groups:
- HEALICOIL™ PK Preloaded Suture Anchors: Participants who have received PEEK Suture Anchor:
  HEALICOIL™ PK Preloaded Suture Anchors
- BIORAPTOR™ 2.3 PK Suture Anchors/BIORAPTOR™ Curved 2.3 PK Suture Anchors: Participants who have received PEEK Suture Anchor:
  BIORAPTOR™ 2.3 PK Suture Anchors/BIORAPTOR™ Curved 2.3 PK Suture Anchors
- MULTIFIX™ S Ultra Knotless Fixation System: Participants who have received PEEK Suture Anchor:
  MULTIFIX™ S Ultra Knotless Fixation System
- FOOTPRINT™ Ultra PK Suture Anchors: Participants who have received PEEK Suture Anchor:
  FOOTPRINT™ Ultra PK Suture Anchors
- TWINFIX™ Ultra PK Suture Anchors/TWINFIX™ Ultra Preloaded and With Needles: Participants who have received PEEK Suture Anchor:
  TWINFIX™ Ultra PK Suture Anchors/TWINFIX™ Ultra Preloaded and with Needles
- SPEEDSCREW™ Knotless Fixation System: Participants who have received PEEK Suture Anchor:
  SPEEDSCREW™ Knotless Fixation System
- SpeedLock Knotless Fixation Device: Participants who have received PEEK Suture Anchor:
  SpeedLock Knotless Fixation Device
Arm/Group | HEALICOIL™ PK Preloaded Suture Anchors | BIORAPTOR™ 2.3 PK Suture Anchors/BIORAPTOR™ Curved 2.3 PK Suture Anchors | MULTIFIX™ S Ultra Knotless Fixation System | FOOTPRINT™ Ultra PK Suture Anchors | TWINFIX™ Ultra PK Suture Anchors/TWINFIX™ Ultra Preloaded and With Needles | SPEEDSCREW™ Knotless Fixation System | SpeedLock Knotless Fixation Device
All-Cause Mortality (participants affected / at risk) | 0/193 | 0/41 | 0/78 | 0/136 | 0/57 | 0/59 | 0/18
Serious Adverse Events (participants affected / at risk) | 15/193 | 7/41 | 13/78 | 10/136 | 1/57 | 4/59 | 0/18
Other Adverse Events (participants affected / at risk) | 40/193 | 27/41 | 38/78 | 24/136 | 5/57 | 4/59 | 0/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HEALICOIL™ PK Preloaded Suture Anchors (N=193) | BIORAPTOR™ 2.3 PK Suture Anchors/BIORAPTOR™ Curved 2.3 PK Suture Anchors (N=41) | MULTIFIX™ S Ultra Knotless Fixation System (N=78) | FOOTPRINT™ Ultra PK Suture Anchors (N=136) | TWINFIX™ Ultra PK Suture Anchors/TWINFIX™ Ultra Preloaded and With Needles (N=57) | SPEEDSCREW™ Knotless Fixation System (N=59) | SpeedLock Knotless Fixation Device (N=18)
ADHESIVE CAPSULITIS IN RIGHT SHOULDER (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unlikely related to device
PULMONARY EMBOLUS (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Unrelated to device
RE-TEAR OF ROTATOR CUFF (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Unrelated to device
RIGHT CARPAL TUNNEL WITH RELEASE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
LEFT SHOULDER RECURRENT ROTATOR CUFF TEAR (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Possibly related to device
R RECURRENT RTC TEAR AND IMPINGEMENT SYNDROME (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Possibly related to device
RECURRENT TEAR OF ROTATOR CUFF WITH NEW TEAR OF THE SUPRASPINATUS AND RECURRENT JOINT IMPINGEMENT (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Possibly related to device
LEFT SHOULDER ADHESIVE CAPSULITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
LEFT SHOULDER PAIN WITH RECURRENT RTC TEAR (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
DECREASED ROM RIGHT SHOULDER (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
RIGHT SHOULDER INCREASE IN PAIN WITH POPPING AND GRINDING, RECURRENT RTC TEAR (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
CONTINUING WEAKNESS RIGHT SHOULDER AND DECREASED ROM (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Possibly related to device
LEFT SHOULDER PAIN AND DECREASED ROM (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
RECURRENT RTC TEAR (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
R SHOULDER INCREASED PAIN, WEAKNESS, LTD. ROM, R RECURRENT RTC TEAR (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Possibly related to device
RIGHT SHOULDER ADHESIVE CAPSULITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Possibly related to device
R SHOULDER SUBACHROMIAL BURSITIS WITH SUPRASPINATOUS TENDINOSIS CAUSING DECREASED MOBILITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Possibly related to device
LEFT SHOULDER PAIN AND WEAKNESS RELATED TO RECURRENT RTC TEAR (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Possibly related to device
RIGHT SHOULDER PAIN, TIGHTNESS AND SPASM WITH PERSISTENT WEAKNESS AND RECURRENT RTC TEAR (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
FELT POP R SHOULDER, DECREASED ROM AND PAIN SINCE, RECURRENT RTC TEAR (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
LEFT SHOULDER SWELLING AND PAIN AFTER PT STRETCH AND RECURRENT LEFT RTC TEAR (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
R SHOULDER PAIN CREPITUS AND STIFFNESS WITH RECURRENT RTC TEAR, (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
RIGHT SHOULDER PAIN AND WEAKNESS, RECURRENT R RTC TEAR, (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
INCREASED PAIN, DECREASED ROM AND WEAKNESS, RECURRENT L RTC TEAR, INSOMNIA R/T PAIN (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
WORSENING LEFT SHOULDER PAIN RADIATING DOWN LEFT ARM, RECURRENT LABRAL TEAR (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
LEFT RTC TEAR, RTC CAPSULE SPRAIN (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
LEFT SHOULDER PAIN WITH DECREASED ROM, STIFF AND SORE, ADHESIVE CAPSULITIS AND RTC TENDONITIS (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
RIGHT SHOULDER PAIN, LTD ROM, RTC TEAR (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
OCCASIONAL LEFT SHOULDER PAIN, STIFFNESS, ADHESIVE CAPSULITIS (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Probable to device
R SHOULDER TENDONITIS, PARTIAL RTC TEAR (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
R SHOULDER ANTERIOR WOUND INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
R SHOULDER PAIN, RECURRENT RTC TEAR (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
R RTC TEAR, TENDONITIS AND WEAKNESS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
CLAVICLE FRACTURE AFTER FALL AT WORK (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Unrelated to device
SPLENIC NECROSIS (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Unrelated to device
PNEMOTHORAX- RIGHT (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — Unrelated to device
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HEALICOIL™ PK Preloaded Suture Anchors (N=193) | BIORAPTOR™ 2.3 PK Suture Anchors/BIORAPTOR™ Curved 2.3 PK Suture Anchors (N=41) | MULTIFIX™ S Ultra Knotless Fixation System (N=78) | FOOTPRINT™ Ultra PK Suture Anchors (N=136) | TWINFIX™ Ultra PK Suture Anchors/TWINFIX™ Ultra Preloaded and With Needles (N=57) | SPEEDSCREW™ Knotless Fixation System (N=59) | SpeedLock Knotless Fixation Device (N=18)
COMPLEX REGIONAL PAIN SYNDROME TYPE II (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unlikely related to device
PAIN ON THE RIGHT SIDE OF HER SHOULDER DOWN HER NECK AND THE MEDIAL BORDER OF HER RIGHT SCAPULA. (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Unrelated to device
RIGHT SIDE ARM PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Unrelated to device
SHOULDER PAIN POST FALL (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — Unrelated to device
LEFT HAND NUMBNESS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
LEFT SHOULDER TENDINITIS/BURSITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unlikely related to device
RIGHT SHOULDER DISCOMFORT SECONDARY TO FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
ADHESIVE CAPSULITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
LEFT SHOULDER ANTERIOR PORTAL REDDENED AND SWOLLEN WITH RESOLVING BICEP ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
RIGHT SHOULDER PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
CONTINUED LEFT SHOULDER WEAKNESS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
ACTIVE RANGE OF MOTION LIMITED BY PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
BICEPS ATROPHY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
SHOOTING PAIN DOWN LEFT ARM (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
RIGHT HAND CONTUSION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
ADHESIVE CAPSULITIS RIGHT SHOULDER (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
INCREASE IN RIGHT SHOULDER PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
NEW ONSET ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
RIGHT ARM LIMITED ROM SECONDARY RIGHT SHOULDER PAIN FROM LIFTING INJURY (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
RIGHT BICEPS TENDONITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
RIGHT SHOULDER ADHESIVE CAPSULITIS POST RCR (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
PAINFUL HERNIATED CERVICAL DISC WITH MYELOPATHY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
BILATERAL SHOULDER PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
LEFT SHOULDER INCREASING PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
LEFT SHOULDER CLICKING, NUMBNESS LEFT ARM, LEFT 4TH AND 5TH FINGERS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
NIGHTMARES FROM PERCOCET (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
INSOMNIA R/T LEFT SHOULDER PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
LEFT SHOULDER PAIN WITH EXERCISING (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
LEFT SHOULDER STIFFNESS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
LEFT SHOULDER SORENESS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
EXACERBATION HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
BICEPS TENDONITIS RIGHT SHOULDER (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
NUMBNESS RIGHT THUMB (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
HERNIATED DISC WITH MYELOPATHY, CONTINUED RIGHT ARM WEAKNESS, RIGHT SCAPULA AREA AND SHOULDER PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
WORSENING RIGHT SHOULDER PAIN AND SWELLING (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
FALL CAUSING RIGHT SHOULDER FORCED ABDUCTION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
RIGHT SHOULDER SORENESS AT TIMES (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
ROTATOR CUFF SPRAIN/STRAIN LEFT SHOULDER (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
INSOMNIA SECONDARY TO RIGHT SHOULDER PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
LEFT HAND THIRD FINGER PARONYCHIA VERY PAINFUL AND TENDER (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
POSTERIOR/LATERAL NUMBNESS RIGHT ARM (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
RIGHT SHOULDER SWELLING (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
PAINFUL ROM (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
RECURRENT 6MM RIGHT RTC TEAR SECONDARY TO DIABETES AND SMOKING CAUSING POOR TISSUE QUALITY (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
INCREASING RIGHT SHOULDER PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
ROTATOR CUFF SPRAIN/STRAIN RIGHT SHOULDER (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
CONTINUING SHOULDER PAIN (General disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
PAIN DOWN ARM TO LEFT HAND 4TH AND 5TH FINGERS (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
LEFT SHOULDER BURSITIS (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
LEFT SHOULDER PAIN WITH DECREASED ROM (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
LEFT SHOULDER PAIN AFTER PT STRENGTHENING EXERCISES (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
LEFT LATERAL EPICONDYLITIS (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
LEFT TRICEPS TENDONITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
TINGLING FROM LEFT ELBOW TO WRIST (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
LEFT ELBOW WARM TO TOUCH WITH DECREASED MOBILITY AND PAIN RADIATING TO WRIST (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
SHOULDER PAIN (General disorders) | 2 (2) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
INCREASED RIGHT SHOULDER PAIN R/T FALL (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
RIGHT SHOULDER INCREASED PAIN AND STIFFNESS R/T CATCHING FALLING CLIENT (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
RIGHT ANKLE SPRAIN WITH SWELLING AND PAIN R/T FALL (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
RIGHT SHOULDER LIMITED ROM AND WEAKNESS (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
INCREASED PAIN RIGHT ANKLE (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
WORSENING PAIN RIGHT SHOULDER (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Possibly related to device
RIGHT SHOULDER IMPINGEMENT SYNDROME, WITH LIMITED ADLS AND NIGHT PAIN (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Possibly related to device
NOCTURNAL AWAKENING DUE TO RIGHT SHOULDER TENDINOSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
RIGHT SHOULDER SWELLING, REDNESS, WARMTH AND PAIN, CELLULITIS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
LEFT SHOULDER PAIN, STIFFNESS, NUMBNESS AND DECREASED SENSATION RELATED TO RECURRENT RTC TEAR (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Possibly related to device
RIGHT SHOULDER ACHING PAIN WITH CERTAIN MOVEMENTS (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
LEFT SHOULDER MILD PAIN AND WEAKNESS (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
DECREASED LEFT SHOULDER STRENGTH (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
LEFT SHOULDER DECREASED ROM AND STRENGTH RELATED RTC RUPTURE (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Possibly related to device
LEFT SHOULDER PAIN WITH DECREASED ROM (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Possibly related to device
LEFT SHOULDER CONSTANT PAIN AND WEAKNESS RELATED TO RECURRENT RTC TEAR (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Possibly related to device
LEFT ARM PAIN BICEP REGION AND LEFT SHOULDER SWELLING (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
SMALL PARTIAL THICKNESS LEFT SUPRASPINATUS TEAR (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
OCCASIONAL SHOULDER PAIN (General disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
NAUSEA AND CONSTIPATION R/T POST-OP OXYCONTIN (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
DISCOMFORT RIGHT BICEP INTO NECK AND DISUSE ATROPHY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
RIGHT SHOULDER PAIN AND WEAKNESS (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
LEFT SHOULDER DULL PAIN AFTER STRENUOUS ACTIVITY (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
INTERMITTENT LEFT SHOULDER PAIN SINCE EXERCISING (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
INTERMITTENT EPISODES OF PERSPIRING AND FEELING OF EXHAUSTION (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
LEFT SHOULDER DECREASED ROM (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
DIVERTICULITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
LEFT SHOULDER WEAKNESS AND PAIN (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
INTERMITTENT LEFT BICEP PAIN AND CRAMPING (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
INCREASED LUE PAIN WITH NUMBNESS AND TINGLING TO LEFT RADIAL DIGITS AND INSOMNIA RELATED TO PAIN (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
INCREASING LEFT SHOULDER PAIN (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
LEFT SHOULDER BURSITIS WITH DECREASED ROM AND WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
THUMB PAIN (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
LEFT SHOULDER PAIN AND RESIDUAL WEAKNESS (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
LEFT SHOULDER PAIN, LTD. ROM, WEAKNESS, DISUSE ATROPHY (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
LEFT RTC SMALL PARTIAL THICKNESS TEAR (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
LEFT SHOULDER STIFFNESS, CONSTANT SORENESS, DECREASED ROM, ACHING AND WEAKNESS (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
RIGHT ANTERIOR SHIN NEURALGIA/SPRAIN (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
MIGRAINE HEADACHES (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
OCCASIONAL DEEP LEFT SHOULDER PAIN (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Possibly related to device
LEFT ARM WEAKNESS (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Possibly related to device
ABDOMINAL PAIN AND CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
L SHOULDER PAIN W/LTD. ROM AND STRENGTH (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
LEFT SHOULDER EDEMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
INCREASED LEFT SHOULDER PAIN, HYPERSENSITIVITY AND PARASTHESIA, QUESTION POSSIBLE RSD (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
CELLULITIS AND PURULENT DRAINAGE LEFT SHOULDER WOUND (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
INTERMITTENT LEFT SHOULDER PAIN (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
RIGHT SHOULDER PAIN WITH DECREASED ROM (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
RIGHT SHOULDER PAIN WITH TIGHTNESS, WEAKNESS, AND DECREASED ROM (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
RECURRENT RTC TEAR (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
INTERMITTENT RIGHT SHOULDER PAIN (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
LEFT SHOULDER ANTERIOR INCISIONS WITH MILD CELLULITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
WORSENING LEFT SHOULDER PAIN AND SWELLING DUE TO FALLING IN SHOWER, CATCHING HERSELF WITH LEFT ARM (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
LEFT SHOULDER STIFFNESS AND LTD. ROM (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
LEFT SHOULDER MILD TENDINOSIS, POSSIBLE SLAP TEAR (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
RIGHT ROTATOR CUFF TENDONITIS, ACJ IMPINGEMENT (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
RIGHT SHOULDER SWELLING AND PAIN (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
LEFT SHOULDER STIFFNESS "SLEPT ON IT WRONG" (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
OCCASIONAL LEFT SHOULDER DECREASED ROM, PAIN, AND WEAKNESS (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
SLIPPED OFF CURB AND FELL ONTO LEFT ARM (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
PAIN FROM LEFT SHOULDER STRAIN (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
RETURNING LEFT SHOULDER PAIN (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unlikely related to device
R SHOULDER PAIN, DECREASED ROM AND BICEPS AREA PAIN (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
RIGHT SHOULDER SURGICAL SCAR SENSITIVITY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
PALPABLE TIGHTNESS RIGHT TRAPEZIUS AREA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
LEFT SHOULDER INTERMITTENT PAIN AND DECREASED ROM (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
CONTINUING RIGHT SHOULDER PAIN AND DECREASED ROM (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
REACHING IN PT AND FELT A "POP" WITH INCREASED PAIN RIGHT SHOULDER (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
RAISED RASH RIGHT FOREARM AND RIGHT ARMPIT (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
NAUSEA FROM PAIN MEDICATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
REDNESS AND SWELLING AROUND INCISION FRONT OF RIGHT SHOULDER (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
RIGHT BICIPITAL GROOVE TENDERNESS AFTER OVERSTRETCHING IN PT (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
WORSENING PAIN RIGHT SHOULDER (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
GLENOHUMERAL INTERNAL ROTATION DEFICIT RIGHT SHOULDER (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
LEFT SHOULDER CONTINUING PAIN (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Possibly related to device
LEFT SHOULDER STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Possibly related to device
WORSENING LEFT SHOULDER PAIN AND DECREASED ROM (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Possibly related to device
LEFT KNEE ARTHROFIBROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
RIGHT SHOULDER PAIN AT NIGHT (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
CONTINUED POST-OP REVISION LEFT SHOULDER PAIN (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
POSSIBLE LEFT CUBITAL TUNNEL SYNDROME (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
LEFT SHOULDER POST. INCISION OPEN W/BLOOD DRAINAGE- SUTURE FELL OUT (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
LEFT SHOULDER WORSENING PAIN, LTD ROM (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
ULNAR NERVE SYMPTOMS AND MEDIAL SCAPULAR PAIN, NECK PAIN (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
HERNIATED DISC WITH MYELOPATHY (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
RECURRING RIGHT ELBOW PAIN, ACUTE RIGHT EPICONDYLITIS (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
L SHOULDER PAIN, DECREASED ROM W/DIFFICULTY SLEEPING @ NIGHT, POSSIBLE ADHESIVE CAPSULITIS (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
LEFT ELBOW PAIN (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
LEFT ELBOW STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
RIGHT FOREARM PAIN AND MUSCLE SPASMS (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
RIGHT SHOULDER INSTABILITY AND PAIN R/T STRAIN/SPRAIN (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
LEFT SHOULDER PAIN POST MUA, LOA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
RECURRENT RIGHT SHOULDER PAIN, POST-OP REVISION (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
RIGHT SHOULDER MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
RIGHT ROTATOR CUFF RE-TEAR (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
ROTATOR CUFF RETEAR (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Unlikely related to device
SEVERE CENTRAL SPINAL STENOSIS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Unrelated to device
HERPES ZOSTER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Unrelated to device
HYPERLIPIDEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Unrelated to device
GENERALIZED ANXIETY DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Unrelated to device
RIGHT ELBOW INJURY, POSSIBLE FRACTURE, OCCURRED DUE TO FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Unrelated to device
MASS OF SOFT TISSUE OF RIGHT UPPER EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Unrelated to device
ADD (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Unrelated to device
HYPERTENSION (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Unrelated to device
INFECTION/SMALL HEMATOMA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to device
ROTATOR CUFF FAILURE / RECURRENT TEAR (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Possibly related to device

LIMITATIONS AND CAVEATS:
No limitations reported

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-01): https://cdn.clinicaltrials.gov/large-docs/67/NCT03826667/Prot_SAP_000.pdf